Official Title of the Study Population-level prevalence, effect on quality of life, and treatment behavior for renal colic and urolithiasis in Poland

Brief Title Renal colic and urolithiasis in Poland

NCT Number NCT06176469

Unique Protocol Id 118.6120.94.2023

Date 06/01/2023

### Questionnaire (aligned with the study protocol)

### R. Demographic parameters:

- R1. Please enter your year of birth:
- R2. Please indicate your sex:
  - 1. Man
  - 2. Woman
- R3. Please indicate your place of residence:
  - 1. City with over 500,000 inhabitants
  - 2. City with 100,000-500,000 inhabitants
  - 3. City with 20,000–100,000 inhabitants
  - 4. City with up to 20,000 inhabitants
  - 5. Rural area
- R4. Please indicate the voivodeship (province) of your residence:
  - 1. dolnośląskie
  - 2. kujawsko-pomorskie
  - 3. lubelskie
  - 4. lubuskie
  - 5. łódzkie
  - 6. małopolskie
  - 7. mazowieckie
  - 8. opolskie
  - 9. podkarpackie
  - 10. podlaskie
  - 11. pomorskie
  - 12. śląskie
  - 13. świętokrzyskie
  - 14. warmińsko-mazurskie
  - 15. wielkopolskie
  - 16. zachodnio-pomorskie
- R5. What is your level of education?
  - 1. Primary
  - 2. Vocational
  - 3. Secondary
  - 4. High

R6. What is your marital status?

- 1. Single
- 2. Married
- 3. Divorced
- 4. Widow/Widower

R7. What is your employment status?

- 1. Employed
- 2. Unemployed
- 3. Retired (pensioner)
- 4. Homekeeper (housewife/husband)

R8. Have you worked or are you currently working in a profession that involves exposure to high ambient temperature (e.g., cooker/baker/miner/steelworker)?

- 1. Yes
- 2. No

R9. Do you or did you have free access to drinking water at work?

- 1. Yes
- 2. No

R10. Do you or did you have free access to a toilet at work?

- 1. Yes
- 2. No

R11. Please select the profession you currently have or had:

- 1. Manual worker
- 2. Scholarly or office worker
- 3. Never been employed

#### **D1-D9. Renal colic-like pain symptoms:**

# SCRIPT: If your answer is "no," proceed to question D10

D1. Have you ever experienced back pain (in the kidney area) that was cramp-like, intermittent, coming and going, and possibly radiating to the groin (commonly referred to as "renal colic")? This pain is typically located along the sides of the back and is unrelated to movement or changes in body position. The pain may also be accompanied by nausea or vomiting.

- 1. Yes
- 2. No

- D2. Did you seek help or treatment for these symptoms?
  - 1. Yes
  - 2. No

### SCRIPT: If your answer is "no," proceed to question D7

- D3. Did you receive help or treatment for these symptoms?
  - 1. Yes
  - 2. No

#### **Multi-answer question**

- D4. What type of treatment did you receive?
  - 1. Over-the-counter medication
  - 2. Prescribed medication
  - 3. Surgical treatment
  - 4. Other
- D5. Are you continuing the treatment that was provided for you?
  - 1. Yes
  - 2. No
- D6. Are you satisfied with the treatment that was provided?
  - 1. Yes
  - 2. No
- D7. Do these symptoms still occur for you, that is, do they recur from time to time?
  - 1. Yes
  - 2. No
- D8. Have the symptoms we are asking about occurred for the first time within the past year, i.e., in the prior 12 months?
  - 1. Yes
  - 2. No
- D9. Which of the following statements best describes your feelings regarding the occurrence of these symptoms?
  - 1. The symptoms generally do not cause me any trouble.
  - 2. The symptoms cause me very little trouble.
  - 3. The symptoms cause me some trouble.
  - 4. The symptoms cause me moderate trouble.
  - 5. The symptoms cause me significant trouble.
  - 6. The symptoms cause me a great deal of serious trouble.

#### **D10-D16. Urolithiasis**

SCRIPT: If your answer is "no," proceed to question D16

D10. Have you ever been diagnosed with urinary tract stones/urolithiasis?

- 1. Yes
- 2. No

#### **Multi-answer question**

D11. Where in the urinary tract was the stone diagnosed?

- 1. Kidney
- 2. Ureter
- 3. Bladder
- 4. I don't know

#### Multi-answer question, answer 4 - deactivates answers 1-3

D12. How was your urinary tract stone diagnosed?

- 1. Ultrasound (USG)
- 2. Computed tomography (CT scan)
- 3. Abdominal X-ray (RTG)
- 4. No additional tests

#### Multi-answer question, answer 8 - deactivates answers 1-7

D13. How was your urinary tract stone treated?

- 1. Observation (without pharmacological or surgical treatment)
- 2. Over-the-counter medication
- 3. Prescribed medication
- 4. Surgical procedure through the urethra (URS)
- 5. Surgical procedure through a puncture in the back (PCNL)
- 6. Surgical procedure through an abdominal incision (open or laparoscopic surgery)
- 7. Stone fragmentation using external shock wave therapy (ESWL)
- 8. Not treated

#### Multi-answer question, answer 5 - deactivates answers 1-4

D14. Was urinary tract stone prevention suggested to you?

- 1. Increased fluid intake
- 2. Dietary changes (dietary recommendations)
- 3. Over-the-counter medication
- 4. Prescribed medication
- 5. No prevention applied

D15. Do you experience recurrent urinary tract stones?

- 1. Yes
- 2. No

D16. Has anyone in your family ever had urinary tract stones? 1. Yes 2. No E. General Health: E1. Please enter your weight in kilograms (approximately): E2. Please enter your height in cm (approximately): |\_|\_| cm Table, singles in row E3. Please indicate which of the following diseases you have and what lifestyle characteristics describe you: **Column list:** 1. Yes 2. No **Rows list:** 1. Hypertension 2. Heart failure 3. Diabetes 4. Gout 5. Liver disease 6. Intestinal disease (e.g., Crohn's disease, fistulas, malabsorption disorders) 7. Chronic kidney disease/Chronic renal failure 8. Hyperparathyroidism 9. Overweight/obesity 10. Polycystic kidney disease 11. Intestinal surgery 12. Sarcoidosis 13. Spinal cord injury 14. Multiple sclerosis 15. Cancer (any) 16. Hematological malignancy (e.g., lymphoma, leukemia, myeloma) 17. Urological malignancy (e.g., prostate cancer, bladder cancer, kidney cancer, ureter cancer, urethral cancer, testicular cancer)

- 18. Benign prostatic enlargement
- 19. Recurrent urinary tract infections
- 20. Neurogenic bladder
- 21. Other urological diseases
- 22. Smoking
- 23. Alcohol consumption (2 or more servings per day)
- 24. Drinking at least 2.5 liters of fluids per day

#### 25. Salting food

#### Table, singles in row

E4. How often do you consume:

#### **Column list:**

- 1. Every day
- 2. Every other day
- 3. Once a week
- 4. Rarely
- 5. Never

#### **Rows list:**

- 1. Beef
- 2. Pork
- 3. Poultry
- 4. Cold cuts, sausages, hot dogs, pâtés, canned food
- 5. Dairy products (e.g., milk, yogurt, eggs, kefir, cheese)
- 6. Cereal products (products made from rye, oats, wheat, corn, rice)
- 7. White bread
- 8. Whole grain bread
- 9. Legumes (e.g., chickpeas, beans, peas, fava beans)
- 10. Soy products
- 11. Fresh fruits
- 12. Fresh vegetables
- 13. Nuts
- 14. Cocoa/chocolate
- 15. Highly processed sweets (e.g., bars, cookies, pastries)
- 16. Spinach
- 17. Strawberries
- 18. Fruit juices
- 19. Sweetened beverages (e.g., soda)
- 20. Coffee
- 21. Tea
- 22. Instant meals/ramen noodles
- 23. Fast food dishes

#### **Table**

- E5. Are you receiving treatment from a urologist?
  - 1. Yes
  - 2. No

- 1. Yes
- 2. No

### E7. Are you receiving treatment from a cardiologist?

- 1. Yes
- 2. No
- E8. Are you receiving treatment from a nephrologist?
  - 1. Yes
  - 2. No
- E9. Are you receiving treatment from a neurologist?
  - 1. Yes
  - 2. No

## **K. International Prostate Symptom Score (IPSS)**

## L. Overactive Bladder-Validated 8-question Screener (OAB-V8)

## Z. General quality of life:

- Z1. If you had to spend the rest of your life in your current general state, how would you describe your well-being?
  - 1. Excellent
  - 2. Satisfied
  - 3. More than half satisfied
  - 4. Half-satisfied
  - 5. Less than half dissatisfied
  - 6. Unhappy
  - 7. Terrible